CLINICAL TRIAL: NCT05113147
Title: Disruptive Behavior in the Operating Room: Systemic Over Individual Determinants
Brief Title: Disruptive Behavior in the Operating Room
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Maria Jesus Lira, Nurse, Pontificia Universidad Catolica de Chile
Other Study IDs: 15-340
Record Dates: First submitted 2021-10-28; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Disruptive Behavior
Keywords: Disruptive Behavior; Patient Safety; Operating Room; Surgeons; Effective Teamwork; Organizational Culture; Qualitative Study
MeSH Terms: conditions — Problem Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: In-depth individual interviews — In-depth individual interviews were based on a semistructured script designed to investigate the perceptions of the participants about the activity they performed, the ideal working conditions, the presence of disruptive behaviors, and their management.

SUMMARY:
Background: The operating room (OR) environment presents specific conditions that put stress on work dynamics. Disruptive behavior (DB) among members of the health team is recognized to affect work dynamics and patient outcomes. The objective was to explore the perceptions of different members of the health team, including surgeons, about the occurrence of DB and the work dynamics in the OR.

Study design: Qualitative exploratory study, based on semi structured individual interviews. Twenty participants were sampled until data saturation, including surgeons, anesthetists, nurses among other. Data extraction from verbatim transcriptions was performed by investigators via qualitative analysis software, using grounded theory framework.

DETAILED DESCRIPTION:
METHODS

A qualitative exploratory study was carried out within an analytical and relational framework of the contents [19,20]. The study was approved by a Scientific Ethics Committee (project ID: 15-340) and meets the quality standards for reporting qualitative Research (COREQ checklist).

Selection of participants Intentional theoretical sampling was performed, which considered the representation of different members of the health team to seek maximum heterogeneity.

The inclusion criterion was that the health members had at least one year of experience in the operating room. Participants were included until achieving data saturation from the information obtained.

Data collection In-depth individual interviews were based on a semistructured script designed to investigate the perceptions of the participants about the activity they performed, the ideal working conditions, the presence of disruptive behaviors, and their management. The final version of the script was reached after the first four interviews. Once the adjustments were made, the same script was used with the other participants.

The interviews were conducted by two interviewers (DZ and MC) with experience in this collection technique and who were not linked to the activities of the health team that was the subject of this study. The information was collected in 2017 and 2018. The participants were invited by email, and once they signed an informed consent, which explained the research´s goal and information about their participation. Once they agreed to participate, the interviewers interviewed an office face-to-face to guarantee privacy and confidentiality. Interviews lasted an average of 45 minutes, and all were audio-recorded and later transcribed verbatim.

Data analysis The participants' responses were analyzed with open and axial coding, based on the grounded theory model to relate the categories emerging from the responses.

Grounded theory is based on the analysis of the narrative contained in the interviews. This in turn leads to the development of codes, categories and themes based on the descriptions to culminate in hypotheses of how these themes interact. Atlas.ti v8.0 software was used for the data analysis (ATLAS.ti Scientific Software Development GmbH, Lietzenburger Str. 75, D-10719 Berlin, Germany).

Six researchers from the team collaborated in the analysis of the transcripts through an iterative process of intersubjective data triangulation sessions until definitive categories and guiding questions were reached regarding the phenomenon under study.

After the analysis, all participants received an email, who explained the findings and asked for feedback (member checking).

ELIGIBILITY:
Inclusion Criteria:

* Health members working in the operating room.

Exclusion Criteria:

* Less than one year of experience in the operating room.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Twenty participants included (surgeons n = 12, anesthetists n = 2, residents n = 2, nurses n = 2, technicians n = 2).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Perceptions about the occurrence of disruptive behaviors and the work dynamics in the operating room | Up to 45 minutes
  In-depth individual interviews were based on a semistructured script designed to investigate the perceptions of the participants about the activity they performed, the ideal working conditions, the presence of disruptive behaviors, and their management

CONTACTS AND LOCATIONS:
Locations (1):
- María-Jesús Lira, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No
To protect the confidentiality of the participants, interview transcripts will not be shared.